CLINICAL TRIAL: NCT03706118
Title: Physiologic Interindividual Variability of Volume and Atrophy in Central Nervous System Structures With Focus on Spinal Cord as Measured by Quantitative Magnetic Resonance Imaging.
Brief Title: Physiologic Volume and Atrophy of Brain and Spinal Cord Measured by Magnetic Resonance Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dana Horakova (Other)
Responsible Party: Sponsor-Investigator, Dana Horakova, Principal Investigator, General University Hospital, Prague
Organization: General University Hospital, Prague (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KHL 182/2017
Record Dates: First submitted 2018-09-17; First posted 2018-10-15 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Cognitive Change; Atrophy Brain; Atrophy; Spinal Cord; Multiple Sclerosis
Keywords: Multiple Sclerosis; Spinal Cord Atrophy
MeSH Terms: conditions — Atrophy; Multiple Sclerosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal, monocentric, interventional study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI and Neuropsychologic testing (Experimental): 102 healthy controls will be examined by magnetic resonance imaging (MRI) of brain, spinal and thoracic cord at month 0, 12, 24 and 36.
  102 healthy controls will be examined by neuropsychological and walking testing designed for patients with multiple sclerosis at month 0, 12, 24 and 36.
  Interventions: Other: Magnetic resonance imaging

INTERVENTIONS:
Other: Magnetic resonance imaging — At month 0, 12, 24 and 36 participants will be examined by quantitative magnetic resonance imaging of brain, cervical and part of thoracic spine.

SUMMARY:
Spinal cord (SC) involvement is prevalent in multiple sclerosis (MS) and contributes importantly to disease progression. To be able reliably evaluate spinal cord volume and its changes in MS patients we need to understand variability of these parameters in sex and age matched healthy controls (HC). To date, no generally available data about these parameters in HC are available.

The objective of this study is to investigate age and sex matched HC by MRI to get the basic set of the data representing both cross sectional values and its longitudinal changes.

The present study will also investigate different strategies how to normalize the absolute spinal cord and brain volume data, what is a relationship between spinal cord volume and brain volume and what is the best protocol to be used in a routine clinical practice.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic immune-mediated inflammatory and neurodegenerative disease that affects central nervous system. Magnetic resonance imaging (MRI) is the main paraclinical examination used to monitor disease activity and response to treatment. However, there is only limited correlation between the clinical symptoms and findings seen on the conventional MRI - a phenomena called clinical-radiological paradox. Measuring whole and regional brain atrophy provides additional information to MRI and seems to correlate better with clinical course and prognosis. In the last two decades, brain atrophy in MS has been exten sively studied, cut-offs for brain volume loss over time has been established and it is likely that it will become an important outcome measure in both clinical studies and routine practice.

Compared to brain atrophy, spinal cord (SC) atrophy and its relation to MS-related disability has been given less attention. This is partly due to technical challenges such as inhomogeneous magnetic field in this region, small physical dimensions of SC and artefacts caused by motion of the SC within the spinal canal together with the flow of cerebrospinal fluid and periodic motion due to respiratory and cardiac cycles. Moreover, focal spinal cord MS lesions may cause both swelling and shrinking of SC that influence its absolute volume, resulting in problems with interpretation of absolute SC volume in MS. Despite all these challenges, it is possible to identify SC lesions and reliably measure SC volume, but there is no "gold standard" (standardized) software for SC volume measurement and no agreement on the SC level (segments) that is most suitable for SC volume loss measurement.

During 2016 we have developed an in-house semiautomatic pipeline for measurement of cervical spinal cord volume that is a part of Scanview program. The segmentation is performed on T2-weighted images. In the first step, a marker is manually placed in a center of an intervertebral disc C3-4 (sagittal plane). Subsequently a cord straightening (manual rotation of the cord to achieve a perpendicular orientation of spinal cord to dorsal part of C3 vertebral body), that enable to reduce partial volume due to the cord orientation. After this centering and straightening,transformation matrix is saved and all subsequent steps are fully automatized. These steps include: 1. Sub-pixel division, 2. Reversing the contrast of T2-weighted images and smoothing by applying a set of median, Gaussian and edge-enhancing filters and 4. Cubic spline interpolation to find a curve that represents a border of a spinal cord with highest probability. Finally, a sum of mean areas of 21 1-mm slices is calculated (1 center slice fixed at center of a intervertebral disc C3-4 and 2 x 10 slices in cranial and caudal direction. Using this new software we have assessed 1,036 MS patients during 2016 and 2017. The intra- and inter-rater variability of SC volume assessment was done by using the intraclass correlation coefficient (ICC) with a two-way mixed absolute agreement and single-measures design. The analysis confirmed very good consistency (> 98%) of the method. The preliminary results showed a significant correlation between spinal cord volume and different clinical phenotypes.

ELIGIBILITY:
Inclusion Criteria:

1. Each participant must provide informed consent in accordance with local regulations
2. Age 18-60 years.

Exclusion Criteria:

1. Not able to undergo MRI examination
2. Not able to be examined 4 times, i.e. M 0, 12, 24, 36 during the next 3 years
3. Pregnancy at the time of enrollment into the study
4. Other disease or medical condition that can influence the volume of brain or spinal cord

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Measure Spinal Cord Volume Change at 12 months during 3 years follow-up in Healthy Controls | Baseline, 12, 24, 36 months
  Evaluation of Magnetic Resonance Imaging from each visit
Measure Spinal Cord Atrophy Change at 12 months during 3 years follow-up in Healthy Controls | Baseline, 12, 24, 36 months
  Evaluation of Magnetic Resonance Imaging from each visit

SECONDARY OUTCOMES:
Measure Whole Brain Volume and Atrophy at 12 months during 3 years follow-up in Healthy Controls | Baseline, 12, 24, 36 months
  Evaluation of Magnetic Resonance Imaging from each visit
Measure Regional Brain Volumes and Atrophies at 12 months during 3 years follow-up in Healthy Controls | Baseline, 12, 24, 36 months
  Evaluation of Magnetic Resonance Imaging from each visit

CONTACTS AND LOCATIONS:
Overall Officials: Dana Horakova, MD, PhD, Principal Investigator — Dpt of Neurology, Charles University and General University Hospital in Prague
Locations (1):
- Dpt of Neurology, Charles University and General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaneckova M, Piredda GF, Andelova M, Krasensky J, Uher T, Srpova B, Havrdova EK, Vodehnalova K, Horakova D, Hilbert T, Marechal B, Fartaria MJ, Ravano V, Kober T. Periventricular gradient of T1 tissue alterations in multiple sclerosis. Neuroimage Clin. 2022;34:103009. doi: 10.1016/j.nicl.2022.103009. Epub 2022 Apr 16. PMID 35561554

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT03706118/Prot_SAP_000.pdf